CLINICAL TRIAL: NCT03639181
Title: A Study to Evaluate the Efficacy and Safety of Genormab Injection in Chinese Patients With Recurrent or Refractory B-cell Non-Hodgkin's Lymphoma (B-NHL)
Brief Title: Clinical Trial in Chinese Patients of B-cell Non-Hodgkin's Lymphoma(GB226)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gxplore-003
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
Keywords: B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB226 3mg/kg every 2 weeks (Experimental): Geptanolimab Injection, 3mg/kg every 2 weeks
  Interventions: Biological: GB226

INTERVENTIONS:
Biological: GB226 — 3mg/kg treat every 2 weeks
  Other Names: Geptanolimab Injection

SUMMARY:
An open-label, single-arm, phase II clinical study of anti-PD-1 antibody GB226 in treatment of recurrent or refractory B-cell non-Hodgkin's lymphoma (B-NHL)

DETAILED DESCRIPTION:
GB226, 3mg/kg/time, is intravenously infused once every two weeks until disease progression, intolerable toxicity or study withdrawal decided by the investigator/subject. It is expected that each subject will be followed for 2 years. Subjects receiving GB226 treatment will be followed once every 2 weeks to the end of this study. If the patients terminate the treatment and their imaging assessment shows no progressive disease (PD), they should be followed once every 6 weeks until progressive disease (imaging evaluation). If the patients have progressive disease (imaging assessment), they should be followed every 3 months until the end of this study or premature withdrawal from the study. Relevant tests and evaluation should be completed at each visit according to standard of care. The follow-up visits can be performed by telephone. During the study, subjects must complete one imaging test and efficacy evaluation every 6 weeks until disease progression. Moreover, patients should be closely monitored for adverse events from subject enrollment to 30 days after the last dosing

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Understanding of procedures and contents of the study, and voluntary signing of written informed consent form;
3. Histopathologically confirmed Primary Mediastinal B-cell Lymphoma (PMBCL):
4. Consent to provide archived tumor tissue samples or fresh tissue samples;
5. ECOG score: 0-1;
6. Expected survival ≥ 3 months;
7. Computed tomography scans performed within 28 days prior to study enrollment should show at least one tumor lesion that can be clearly measured in two perpendicular directions. The longest diameter of intranodal lesion is >1.5 cm, and the longest diameter of extranodal lesion is >1.0 cm (according to the 2014 lugano standard);
8. Blood routine requirements: hemoglobin ≥80 g/L, neutrophil ≥1.0 × 109 /L, platelet ≥75× 109 /L (before test)No blood transfusion or biostimulant for 14 days);
9. Serum creatinine ≤1.5 ULN or creatinine clearance ≥50 mL/min (Cockcroft-Gault formula)
10. Total bilirubin ≤1.5 ULN (Gilbert syndrome allows ≤5 ULN), aspartic acid transaminase (AST)ALT≤ 2.5 ULN (AST and/or ALT≤5×ULN is allowed in patients with liver metastasis)
11. Thyroid function indexes: thyrotropic hormone (TSH) and free thyroxine (FT3/FT4) were in the normal range.If TSH and FT3 are not in the normal range, FT4 can be included.
12. Women should be confirmed not pregnant within 7 days before administration; both males and females agree to do effective contraceptive measures during the trial and 6 months after completion;
13. Patients were able to visit according to the schedule and communicate well with the investigator and complete the study in accordance with the protocol

Exclusion Criteria:

1. Patients with history of other malignant tumors (except cured cervical cancer in situ, basal cell carcinoma or squamous epithelial cancer) may not participate in the study unless complete response lasts for at least 2 years prior to enrollment, and it is estimated that no other treatment will be required throughout the study;
2. Definite central nervous system (CNS) infiltration of lymphoma, including brain parenchyma, meningeal invasion or spinal cord compression;
3. Systemic chemotherapy and targeted therapy were carried out within 2 weeks before the experimental medication, and radical/generalized radiotherapy was carried out within 4 weeks.Anti-tumor biotherapy (tumor vaccine, cytokines or growth factors for the purpose of tumor control); In 1 weeksLocal palliative radiotherapy;
4. A systemic corticosteroid (prednisone >10 mg/ d or equivalent) was administered within 2 weeks before administration;
5. Autologous hematopoietic stem cell transplantation was performed within 2 months and allogeneic hematopoietic stem cell transplantation was performed within 5 years plant;
6. Major surgery under general anesthesia was performed within 4 weeks before the trial. Local anesthesia/epidural anesthesia within 2 weeks surgery
7. Active, known history of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, and type iiRheumatoid arthritis, inflammatory bowel disease, hashimoto's thyroiditis, etc., except: type 1 diabetes, only through hormonesHypothyroidism that can be controlled with alternative therapies, skin diseases that do not require systemic treatment (e.g. vitiligo, psoriasis),Controlled celiac disease or disease in which no recurrence is expected without an external stimulus
8. Uncontrolled hypertension (systolic blood pressure > 140mmHg and/or diastolic blood pressure > 90mmHg) or pulmonary hypertension orUnstable angina pectoris; Had myocardial infarction or bypass or stent surgery within 6 months before the drug administration; Meet in New YorkA history of chronic heart failure at NYHA level 3-4; Valvular disease with clinical significance; Need to beTreated severe arrhythmia (except atrial fibrillation and paroxysmal supraventricular tachycardia), including QTc interphase male ≥450ms, female ≥470ms (calculated by Fridericia formula); Left ventricular ejection fraction (LVEF) < 50%;Cerebrovascular accident (CVA) or transient ischemic attack (TIA) etc. occurred within 6 months before the administration;
9. Other serious medical conditions, including but not limited to: uncontrolled diabetes, active digestive tract ulcers,Active hemorrhage, etc;
10. Active infectious persons requiring systemic treatment;
11. Previous or current active TB infectious patient;
12. Human immunodeficiency virus antibody (hiv-ab) and treponema pallidum antibody (tp-ab) were positive. Hepatitis c antibody (HCV-Ab) positive, and the upper limit of normal value of HCV RNA quantitative > detection unit; Hepatitis b virus surface antigen (HBsAg)Positive, and HBV DNA quantitative > detection unit normal limit;
13. Complications that require systemic immunosuppressive drug therapy or that require an immunosuppressive dose (prednisone)> 10 mg/ day or equivalent dose of similar drugs) systemic treatment complications; In the absence of active autoimmune diseaseIn this case, inhaled or locally administered steroids and > 10mg/ d prednisone or equivalent dose are allowed;
14. Adverse reactions from previous treatment did not return to level 1 or below before medication (CTCAE5.0) (alopecia and chemotherapyDrug induced grade 2 neurotoxicity excepted);
15. Uncontrolled or symptomatic pleural or pericardial effusion;
16. Previous use of anti-pd-1 antibodies, anti-pd-l1 antibodies, anti-pd-l2 antibodies or anti-ctla-4 antibodies (orAny other antibodies that act on T cell synergistic stimulation or checkpoint pathways);
17. Other experimental drugs or experimental instruments were used within 30 days before administration;
18. Live or attenuated vaccines were administered within 4 weeks of trial administration;
19. A history of drug abuse or drug abuse was enquired;
20. History of interstitial lung disease;
21. Lactating women who do not want to stop breastfeeding;
22. Known allergy to recombinant humanized pd-1 monoclonal antibody or any of its excipients; A known history of allergic disease or severe allergies;
23. Patients with insufficient communication, understanding and cooperation, or poor compliance, can not be guaranteed to follow the program requirements;
24. The researchers concluded that participants in this clinical trial were not suitable for a variety of other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | up to 52 weeks
  To evaluate the efficacy of GB226 as defined by objective response rate, in patients with B-NHL.

SECONDARY OUTCOMES:
Duration of response, DOR | up to 52 weeks
  To evaluate the duration of response (DOR) of GB242 in patients with B-NHL.
Overall survival, OS | up to 52 weeks
  To evaluate the duration from the first administration to death because of any reason in patients with B-NHL.
Progression-free survival, PFS | up to 52 weeks
  To evaluate the efficacy of GB226 as defined by progression-free survival, in patients with B-NHL.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No